CLINICAL TRIAL: NCT05256472
Title: Phase II Trial of Cadonilimab (AK104) Monotherapy or AK104 Plus Axitinib in Advanced/Metastatic Renal Cell Carcinoma (RCC)
Brief Title: A Study of AK104 Monotherapy or AK104 Plus Axitinib in Advanced/Metastatic Renal Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-213
Record Dates: First submitted 2022-01-24; First posted 2022-02-25 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Renal Cell Carcinoma; First-line Treatment
Keywords: AK104; Axitinib
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Axitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK104 monotherapy cohort (Part 1) (Experimental): Subjects in this cohort will randomly receive three different dosage of AK104 monotherapy administered intravenously.
  Interventions: Drug: AK104
- combination treatment cohort (Part 2) (Experimental): Subjects in this cohort will receive AK104 (RP2D, administered intravenously) plus Axitinib 5 mg bid, administered orally.
  Interventions: Drug: AK104; Drug: axitinib

INTERVENTIONS:
Drug: AK104 — anti-PD-1/CTLA-4 bi-specific antibody drug; RP2D intravenously (IV)
Drug: axitinib — an oral, small molecule, TKI selective for VEGFRs 1, 2 and 3; 5mg bid orally
  Arms: combination treatment cohort (Part 2)

SUMMARY:
This is a Phase II, open-label trial to evaluate the efficacy and safety of AK104 monotherapy or AK104 in combination with axitinib as a first-line treatment for advanced/metastatic renal cell carcinoma (RCC). There are two parts in this trial. In part 1 of this study, subjects with unresectable advanced clear cell or non-clear cell renal cell carcinoma (ccRCC or nccRCC) who had not received systemic therapy for advanced disease will be enrolled to randomly received three different dosage of AK104 monotherapy. In part 2 of this study, subjects with unresectable advanced clear cell renal cell carcinoma (ccRCC) who had not received systemic therapy for advanced disease will be enrolled to receive AK104 plus Axitinib. All subjects will receive treatment until disease progression, development of unacceptable toxicity, death, a decision by the physician or patient to withdraw from the trial. The primary endpoint is ORR per RECIST v1.1 as assessed by investigators.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent/assent for the trial.
2. Be≥18 and ≤ 75 years of age on day of signing informed consent, no matter male or female.
3. Have Karnofsky performance status (KPS) ≥ 70% as assessed within 10 days prior to first dosing of AK104.
4. Have estimated life expectancy of at least 3 months.
5. Have histologically or cytologically confirmed diagnosis of RCC with advanced/metastatic disease (i.e., Stage IV RCC per American Joint Committee on Cancer) with clear cell or non-clear cell component (part 1) or solely clear cell component (part 2).
6. Have received no prior systemic therapy for advanced RCC . Note: Prior neoadjuvant/adjuvant therapies are acceptable if disease progression occurred > 12 months after last dosage of neoadjuvant/adjuvant treatment.
7. Have measurable disease per RECIST 1.1 as assessed by the investigator /site radiologist. (brain metastases were excluded).
8. Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides.
9. Adequate organ function as determined by:

   1. Hematology: i. absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L (1,500/mm3); ii. platelets ≥ 100 × 10^9/L (100,000/mm3); iii. hemoglobin ≥ 90 g/L.
   2. Renal: i. calculated creatinine clearance * (CrCl) ≥ 50 mL/min; * CrCl will be calculated using the Cockcroft-Gault formula CrCL (mL/min) = {(140-age) × body weight (kg) × F }/(SCr (mg/dL) × 72) Where F = 1 for males and F = 0.85 for females; SCr = serum creatinine. ii. urine protein < 2 + or 24-hour urine protein must be < 2.0 g.
   3. Hepatic: i. serum total bilirubin (TBil) ≤ 1.5 × ULN; ii. AST and ALT ≤ 2.5 × ULN, ≤ 3.0 × ULN with liver metastasis; iii. serum albumin (ALB) ≥ 28 g/L.
   4. Coagulation function: i. international normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.
   5. Cardiac Function: i. Left ventricular ejection fraction (LVEF) ≥ 50%.

Exclusion Criteria:

1. Has a known additional malignancy that has progressed or has required active treatment in the last 3 years. Note: Subjects with basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or carcinoma in situ are not excluded.
2. Has had prior treatment with any anti-PD-1, or PD-L1, or PD-L2 agent or an antibody targeting any other immune-regulatory receptors or mechanisms. Examples of such antibodies include (but are not limited to) antibodies against IDO, IL-2R, GITR，CTLA-4，CD40, CD137.
3. Has received prior therapy with VEGF/VEGFR or mTOR targeting agents.
4. Has received radiotherapy within 14 days prior to start of study treatment and has not recovered adequately from any toxicity and/or complications from prior radiotherapy.
5. Has newly diagnosed brain metastases or known symptomatic brain metastases requiring steroids. Subjects with previously diagnosed brain metastases are eligible if they have completed their treatment and have recovered from the acute effects of radiation therapy or surgery prior to receiving first dose of trial treatment, have discontinued corticosteroid treatment for these metastases for at least 3 days and are neurologically stable.
6. Had major surgery 4 weeks or major radiation therapy 2 weeks prior to receiving first dose of trial treatment. Prior palliative radiotherapy to metastatic lesion(s) is permitted, provided it has been completed at least 48 hours prior to receiving first dose of trial treatment.
7. Has active autoimmune disease that might deteriorate when receiving an immunostimulatory agents. Subjects with diabetes type I, vitiligo, psoriasis, hypo-or hyperthyroid disease not requiring immunosuppressive treatment are eligible.
8. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to receiving first dose of trial treatment.
9. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
10. Has an active tuberculosis and syphilitic infection.
11. Has a known history of Human Immunodeficiency Virus (HIV) infection (HIV antibodies).
12. Has known active Hepatitis B (e.g., Hepatitis B surface antigen [HBsAg] reactive and HBV-DNA>200 IU/ml) or Hepatitis C virus (e.g., HCV RNA [qualitative] is detected).
13. Has poorly controlled hypertension defined as systolic blood pressure (SBP) ≥ 140 mm Hg and/or diastolic blood pressure (DBP) ≥ 90 mmHg.
14. Has active bleeding disorder or other history of significant bleeding episodes within 30 days of screening.
15. Has been pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment (30 days for axitinib, whichever occurs last).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-22 (Estimated)

PRIMARY OUTCOMES:
ORR per RECIST v1.1 as assessed by investigators | Up to 2 years
  ORR is the proportion of subjects with complete response(CR) or partial response(PR) , based on RECIST v1.1

SECONDARY OUTCOMES:
Deep response rate | Up to 2 years
  (% patients with >75% tumor reduction at 6 months ) per RECIST v1.1
Duration of response (DOR) | Up to 2 years
  Duration of response (DOR) assessed according to RECIST v1.1
Disease control rate (DCR) | Up to 2 years
  Disease control rate (DCR) assessed according to RECIST v1.1
Progression-free survival (PFS) | Up to 2 years
  PFS is defined as the time from the the start of treatment till the first documentation of disease progression (per RECIST v1.1 criteria) assessed by the investigator or death due to any cause (whichever occurs first).
Overall survival (OS) | Up to 2 years
  Overall survival is defined as the time from the start of treatment until death due to any cause.
Peak Plasma Concentration (Cmax) | Up to 2 years
  The maximum (or peak) plasma concentration of AK104 in subjects treated with AK104 plus axitinib.
Area under the plasma concentration versus time curve (AUC) | Up to 2 years
  AUC = Area under the plasma concentration of AK104-time curve. The area under the plasma concentration time curve (AUC) is a measure of overall exposure to the drug
Immunogenicity assessment | Up to 2 years
  Number and percentage of subjects with detectable anti-drug antibodies (ADAs) treated with AK104 plus axitinib

CONTACTS AND LOCATIONS:
Overall Officials: Dingwei Ye, MD, Principal Investigator — Shanghai Cancer Center of Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No